CLINICAL TRIAL: NCT03224039
Title: Comparison of Intranasal Sufentanil Versus Intravenous Morphine for the Management of Acute Pain
Brief Title: Intranasal Sufentanil Versus Intravenous Morphine for the Management of Acute Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Brooklyn Hospital Center (Other)
Responsible Party: Principal Investigator, Billy Sin, Director, Emergency Medicine Clinical Research Program, The Brooklyn Hospital Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 954045-5
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Sufentanil; Saline Solution; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Assignment of treatment will be based on randomization. Each patient will be assigned a study number that would correspond to a specific treatment. Only the primary investigator (B.Sin) and the pharmacist procuring the study intervention will be unblinded to the treatment. The physician, nurse, research associate responsible for collecting data, and independent biostatistician responsible for interpreting the data will be blinded. Assignment of treatment will be placed in a opaque envelope where it would be opened only by the pharmacist will who be procuring the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal sufentanil (Experimental): Treatment arm to include
  1. Sufentanil 0.7 mcg/kg intranasal (IN) x 1 dose
  2. Normal saline 1ml intravenous (IV) push x 1 dose
  Interventions: Drug: Sufentanil; Drug: Normal saline
- Intravenous morphine (Active Comparator): b. Treatment B:
  1. Normal saline 0.3 mL IN x 1 dose
  2. Morphine 0.1 mg/kg IV push x 1 dose
  Interventions: Drug: Normal saline; Drug: Morphine

INTERVENTIONS:
Drug: Sufentanil — Intranasal for one dose (experimental)
  Arms: Intranasal sufentanil
Drug: Normal saline — Intravenous for one dose as placebo (to be administered with sufentanil or morphine arm as part of double-blinding). If patients are randomized to receive IN sufentanil, they will also receive IV normal saline. If patients are randomized to receive IV morphine, they will also receive IN normal saline.
Drug: Morphine — intravenous push for one dose (active comparator)
  Arms: Intravenous morphine

SUMMARY:
This study will be a single-center, randomized, controlled trial conducted in the Brooklyn Hospital Center's Emergency Department (ED) expected to last 2 years. The sample size will be 40 patients with 20 patients in each treatment arm.

The data points to be collected in the study are as follows: baseline characteristics (baseline pain score, date of birth, age, gender, weight and ethnicity), NRS pain scores at 5, 10, 20, and 30 minutes, dose of study treatment administered, incidence of adverse effects, time to patient discharge following administration of study treatment, patient satisfaction of pain control based on a 10-point Likert Scale, number of patients who required rescue analgesia, and amount of rescue analgesia required. 4.

Once informed consent is obtained, patients will be randomized to receive Treatment A (sufentanil 0.7 mcg/kg intranasally (IN) and normal saline 1ml IV push) OR Treatment B (Normal saline 0.6 mL IN and morphine 0.1 mg/kg IV push). It should be noted that during the study period, use of additional morphine or adjuvant analgesics outside of the designated time intervals is allowed. The decision to use adjuvant analgesics is the decision of the attending physician assigned to the patient in the Emergency Department (ED).

DETAILED DESCRIPTION:
This study will be a single-center, randomized, controlled trial conducted in the Brooklyn Hospital Center's Emergency Department (ED)

Intervention:

Study participants will be randomized to receive one of the two study treatments below:

1. Treatment A:

   1. Sufentanil 0.7 mcg/kg IN x 1dose (max of 1 mL administered per nostril)
   2. Normal saline 1ml IV push x 1dose
2. Treatment B:

   1. Normal saline 0.3 mL IN x 1 dose
   2. Morphine 0.1 mg/kg IV push x 1dose
3. Rescue protocol:

Regardless of assignment to Treatment A or Treatment B, if severity of pain is ≥ 5 on the NRS, IV morphine dosed at 0.1 mg/kg IV push (max dose: 10 mg) may be administered at the discretion of the attending physician or medical resident assigned to the patient at designated intervals (5, 10, 20, and 30 minutes after administration of study treatment)

Process

1. Identification of patients with chief complaints or visit reasons of "acute pain", "musculoskeletal pain", "back pain", "abdominal pain", "fracture", "headache", "lacerations", and "sprains" via the Emergency Department's Status board by Research Associate (RA) or study investigators
2. Screening of potentially eligible patients with inclusion/exclusion criteria checklist via chart review by RA or study investigators.
3. If patient is eligible, the RA or study investigators will approach the medical resident or attending physician to confirm if the patient's visit reason is acute pain. If a medical decision is made by the attending or resident to treat the patient for acute pain, the RA (along with the medical resident, with approval from the attending physician) or study investigators will approach the patient to obtain informed consent and explain potential risks and benefits associated with receiving study interventions. Only study investigators will sign informed consent forms as per IRB protocol.
4. Once informed consent is obtained, patients will be randomized to receive Treatment A (sufentanil 0.7 mcg/kg intranasally (IN) and normal saline 1ml IV push) OR Treatment B (Normal saline 0.6 mL IN and morphine 0.1 mg/kg IV push). It should be noted that during the study period, use of additional morphine or adjuvant analgesics outside of the designated time intervals is allowed. The decision to use adjuvant analgesics is the decision of the attending physician assigned to the patient in the Emergency Department (ED).
5. Order will be placed in the electronic medical record (EMR) by the medical resident, attending physician, or pharmacist under the permission of the attending physician for a study intervention.
6. Upon receiving the medication order in the EMR, the order will be verified by the pharmacy. The pharmacy will then prepare either a sufentanil IN syringe and placebo injection or morphine injection and placebo IN syringe based on the study number assigned to the patient. The study investigators or RA assigned to the study will obtain the medication preparations from the pharmacy. Medication preparations will only be labeled with patient number and study number. No other identifying markers will be placed on the labels.
7. The nurse assigned to the patient or physician from the research team will administer the intervention medications. During administration of the intervention, the patient will be connected to a cardiac monitor for monitoring of possible cardiovascular adverse events.
8. An RA or study investigator will approach the patient to assess and record primary outcomes and secondary outcomes at designated time intervals. The data will be recorded on paper data collection sheets (see attached forms). The primary study investigator will not take part in data collection or analyses. If additional analgesic medications are requested by the patient, the orders will be placed by the medical resident or attending physician assigned to the patient.
9. All data collected on the paper data collection sheets will be transcribed into an encrypted and password protected electronic database by the RA. All patient identifiers will be de-identified in the database and all participants will be assigned a study participant number. This database will be stored on ED computers only and only RA's and study investigators will have access to it. The paper data collection sheets will be stored in a stationary, locked cabinet in the ED for safe keeping. At the end of the study, these records will be maintained according to the hospital's record-retention policy.
10. At the conclusion of study enrollment, an independent biostatistician will analyze the data. Only data from patients with diagnoses relating to acute pain and completed the study protocol without use of rescue analgesia during the designated time will be included in the study. Once the initial data analysis is complete, the log which details whether study participants received sufentanil IN or morphine IV will be revealed to the biostatistician for final data analysis and compilation.
11. At the conclusion of the study, final results and conclusions will be presented to the IRB. All data recorded on the paper data collection sheets will be destroyed and all data on the electronic databases will be deleted.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* presenting to emergency department (ED) with chief complaint of acute generalized pain (including abdominal pain, headache, musculoskeletal pain, back pain, flank pain, joint sprains, lacerations, and fractures) with onset of within 6 hours
* pain score of 5 or greater on numerical pain scale (NRS)
* provides informed consent

Exclusion Criteria:

* reported or documented allergy to sufentanil, morphine, fentanyl, alfentanil, remifentanil, hydrocodone, codeine, hydromorphone, levorphanol, oxycodone, or oxymorphone,
* hemodynamic instability (defined as heart rate not within 60-110bpm
* respiratory rate not within 12-20 bpm
* blood pressure not within 90/50-180/100
* oxygen saturation not within 94-100%)
* refuse to provide "informed consent" form
* nasal obstruction/congestion
* complaint of chest pain
* recent head trauma/injury
* past medical history of hepatic impairment (including history of transplant), renal impairment or chronic renal disease (including history of transplant), chronic alcohol abuse, respiratory disease (ie. hypoxia, hypercapnia, COPD),
* seizure disorder
* thyroid disorders
* language barrier or inability to effectively communicate pain
* weighing > 140 kg
* pregnancy
* active breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-01; Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain score | 10 minutes after initiation of study intervention
  10 point Numeric Rating Scale will be used to assess pain

SECONDARY OUTCOMES:
Adverse events | throughout study period (30 minutes)
  Incidence of adverse events in each group
Mean dose of rescue analgesia required | throughout study period (30 minutes)
  average dose of rescue analgesia required for both groups
Patient satisfaction scores | throughout study period (30 minutes)
  10 point (1-lowest, 10-highest) scores will be used
Number of patients who required rescue analgesia | throughout study period (30 minutes)
  number of patients within each group
Length of stay | throughout study period (30 minutes)
  ED length of study for each group

CONTACTS AND LOCATIONS:
Locations (1):
- The Brooklyn Hospital Center, Brooklyn, New York, United States